CLINICAL TRIAL: NCT03197545
Title: Determining the Risk of Stress Fracture in IDF Soldiers Based on SNPs Identified for Osteoporosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Collaborators: Bar-Ilan University, Israel (Other)
Responsible Party: Principal Investigator, YEHUDA DAVID, Principal Investigator, Medical Corps, Israel Defense Force
Other Study IDs: 1579-2015
Record Dates: First submitted 2017-06-19; First posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Stress Fracture
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA samples will be taken by a sample of the patient's saliva from the inside of the cheek by a sterile specific kit designed for the preservation and subsequent production of DNA from the kit (FTA card).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Stress fracture group: 110 recruits diagnosed (clinicaly and/or by imaging) with at least one stress fracture, during basic and advanced infantry trainig.
- Traumatic fracture group: 110 infantry recruits with medical history of having at least one traumatic fracture, during their life (from birth up to date).
- Control group: 220 healthy infantry recruits never diagnosed with stress fracture or traumatic fractures

SUMMARY:
The study is a genetic historical cohort study in a military combat recruits - this study does not examine a specific treatment but rather examines a statistical link between medical history of traumatic fractures, clinical diagnosis of stress fractures and the presence of unique SNPs in subjects DNA.

DETAILED DESCRIPTION:
Finding a statistically significant correlation between SNPs associated with BMD - Osteoporosis, with recruits who were diagnosed with Stress Fractures during basic and advanced infantry training. Greatest importance will be shown in the power calculation: we suggest that the P-value threshold value of the selected SNPs be adjusted downwards to a lower threshold of P <1.0x10-3 (i.e. equal to 50 independent tests).

We will examine the presence or absence of 96 SNPs - 76 SNPs that were previously validated as significant with low BMD or Osteoporosis and 20 SNPs offered for Stress Fractures with recruits who were diagnosed with Stress Fractures during basic training (basic training lasts four months - six months) using SNP Genotyping Analysis-TaqMan Assays. The buccal swab will be taken from recruits who served for at least four months and up to six months in the IDF - Infantry Corps. Buccal swabs will be taken at a single meeting from recruits serving between 4 and 6 months in the IDF - Infantry Corps, which will be used to compare using SNP Genotyping Analysis-TaqMan Assays with the SNPs listed above. In addition, in this single meeting, the recruits will fill out a questionnaire in which they will be asked whether they experienced traumatic fracture from their youth to the time of filling the questionnaire (recruits who experienced traumatic fractures but are not diagnosed with stress fractures constitute as a control group in the research).

There will be one meeting with recruiters who served for at least four months and up to six months in the IDF - infantry. At this meeting, the recruits will be sampled with a buccal swab and fill out a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* All participants (440) in the research are male.
* All participants (440) are recruits who serve 4-6 months in the IDF - infantry - basic training.
* 110 recruits with a stress fracture diagnosis in their medical portfolio.
* 110 recruits who have Section 4161x flaw (section Eclipse: a long bone fracture)
* 220 recruits without the aforementioned impairment clause and the above mentioned diagnosis (referred as control group).

Exclusion Criteria:

* Recruit who left the unit before conducting the research.
* A recruiter who did not complete his training due to a course that lasted over two weeks while carrying out basic training.
* A recruiter who did not complete his basic training due to absenteeism.
* A recruiter who has not completed his basic training due to problems with the service conditions.
* A recruiter who has not completed his basic training due to the reduction of a medical profile.
* A recruiter who did not complete his basic training due to a decrease in the recruitment cycle.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 440 male infantry recruits training in an IDF (the Israel Defense Forces) boot camp in Israel
Sampling Method: Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Finding a statistically significant correlation between SNPs associated with BMD - Osteoporosis, with recruits who were diagnosed with Stress Fractures during basic and advanced infantry training. | There will be one meeting with recruiters who served for at least four months and up to six months in the IDF - infantry. At this meeting, the recruits will be sampled with a buccal swab and fill out a questionnaire.
  We will examine the presence or absence of 96 SNPs - 76 SNPs that were previously validated as significant with low BMD or Osteoporosis and 20 SNPs offered for Stress Fractures with recruits who were diagnosed with Stress Fractures during basic training (basic training lasts four months - six months) using SNP Genotyping Analysis-TaqMan Assays. The buccal swab will be taken from recruits who served for at least four months and up to six months in the IDF - Infantry Corps. Buccal swabs will be taken at a single meeting from recruits serving between 4 and 6 months in the IDF - Infantry Corps

CONTACTS AND LOCATIONS:
Overall Officials: Izhak Haviv, Prof., Study Chair — Bar-Ilan Faculty of Medicine, Safed; David Karasik, Prof., Study Director — Bar-Ilan Faculty of Medicine, Safed
Locations (1):
- Bar Ilan University, Safed, Israel

IPD SHARING:
Plan to Share IPD: No
Data will be published after statistical analysis only.